CLINICAL TRIAL: NCT07025356
Title: Combined Minimally Invasive Vagal Cranial Nerve and Trigeminocervical Complex Peripheral Nerve Stimulation In Severe Painful Peripheral Neuropathy
Brief Title: Observational Study of the the Use of a Trigeminal Vagal Nerve Stimulator in the Routine Care of Native Americans With Diabetic Neuropathy Pain. Pain Scores, Drug Use and Glucose Measurements Will be Assessed
Status: Completed | Type: Observational
Sponsor: Vagus Nerve Society (Other)
Responsible Party: Sponsor
Other Study IDs: VNS 001
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Neuropathy With Neurologic Complication
Keywords: Vagus; diabetic neuropathy; auricular; stimulation
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Native Americans with Diabetic Neuropathy Pain: Use of Trigeminal Vagus cervical nerve stimulation for diabetic neuropathy pain
  Interventions: Drug: Implantation of a trigeminal Vagus cervical nerve stimulator system; Device: Implantation of a neurostimulator system for trigeminal vagal cervical nerve stimulation

INTERVENTIONS:
Drug: Implantation of a trigeminal Vagus cervical nerve stimulator system — The NS 100 is a medical device used for the treatment of diabetic neuropathy pain. Routine observational monitoring will be performed
Device: Implantation of a neurostimulator system for trigeminal vagal cervical nerve stimulation — The medium term outcomes of neurostimulation will be assessed on diabetic neuropathy pain, glucose and drug usage

SUMMARY:
This is an observational study that will follow patients in the course of routine care and measure pain levels, glucose assessments and drug utilization for native American patients with diabetic neuropathy

DETAILED DESCRIPTION:
Patients with diabetic neuropathy pain will have an NS100 device implanted for chronic diabetic neuropathy pain consistent with onlabel indication. All patients will be followed for 90 days post implant to measure improvements in pain, drug utilization and glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Neuropathy Pain History of failed treatment WIlling to follow blood glucose and pain scores for 90 days

Exclusion Criteria

* Bleeding diathesis Pregnancy Cardiac monitoring device Implantable Neurostimulator Inability to give informed consedn

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Native American Population with Diabetic Neuropathy pain
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain scores over time | 90 days
  Periodic pain scores will be measured for 90 days and possibly longer

SECONDARY OUTCOMES:
glucose levels will be measured over time | 90 days
  Serum glucose levels will be followed on patients receiving neurostimulation

CONTACTS AND LOCATIONS:
Overall Officials: Claire Marie Rangon, MD PHD, Study Director — Vagus Nerve Society
Locations (1):
- Continuum of Care Clinic, Pine Ridge, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
Want to maintain patient autonomy